CLINICAL TRIAL: NCT00773136
Title: Effect of Bimatoprost (Lumigan) in Gel Suspension Applied to the Eyelashes on Eyelash Growth
Brief Title: Eyelash Growth From Application of Bimatoprost in Gel Suspension to the Base of the Eyelashes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Sara T. Wester, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 20070706
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Hypertrichosis
Keywords: Bimatoprost; Eyelash lengthening; Prostaglandin Analogs; Cosmetics
MeSH Terms: conditions — Hypertrichosis | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bimatoprost Suspension (Active Comparator): Intervention to be administered: Each subject was given two suspensions, one mixed with Bimatoprost and one mixed with normal saline. They were instructed to use each suspension to a pre-determined eyelash (prepared prior to study enrollment in double blind fashion and marked after randomization with right and left). The intervention was the one eye with the Bimatoprost.
  Interventions: Drug: Bimatoprost Suspension

INTERVENTIONS:
Drug: Bimatoprost Suspension — see prior
  Other Names: Lumigan

SUMMARY:
Objective: To determine if Lumigan (bimatoprost) causes increased lash length when used in gel suspension applied to the base of the eyelashes. Methods: Subjects recruited from the Bascom Palmer Eye Institute were screened and those who met inclusion criteria were enrolled. Each participant received two vials of gel suspension, which contained bimatoprost and normal saline, respectively, each mixed 1:1 with GonakTM gel and labeled "right eye" and "left eye" according to randomization. The suspension was applied to the eyelashes every evening on the designated eye for 6 weeks. Lash length was measured with a caliper at enrollment, at weekly intervals during the study and at 1 and 3 months after study completion. Visual acuity, ocular symptoms, intraocular pressure and photographs were documented at these same intervals. Results: The average eyelash growth in the Lumigan group was 2.01mm (vs. control average of 1.13mm) which was a statistically significant difference (p=0.009). The average intraocular pressure decreased equally in both groups (2.14 mmHg). No change in visual acuity or iris discoloration was noted in any of the subjects. Discussion: Our data showed an increase in eyelash length with use of Lumigan in gel suspension, suggesting that it may have eyelash lengthening properties.

DETAILED DESCRIPTION:
Study completed

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 20 and less than 90 and patients who have previously used and are comfortable with applying mascara.

Exclusion Criteria:

* History of glaucoma, uveitis, pregnancy, allergic reaction to prostaglandins or the gel suspension, alopecia, and previous usage of other eyelash growth enhancement.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy W Lee, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Bascom Palmer Eye Institute, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Through study advertisement with IRB approved flyers at the Bascom Palmer Eye Institute, 23 subjects were recruited for initial evaluation. Study recruitment and enrollment began in February 2008 and the study was completed in July of 2008, including 3 month post suspension use evaluations.
Groups:
- Bimatoprost Mixed With Gonak Into a Gel Suspension: Each subject was given two suspensions, one of Bimatoprost mixed with Gonak into a gel suspension and one with Gonak mixed with normal saline. They were instructed to use each suspension to a pre-determined eyelash (prepared prior to study enrollment in double blind fashion and marked after randomization with right and left). The solution vials were labeled right or left eye.
Period: Overall Study
Arm/Group | Bimatoprost Mixed With Gonak Into a Gel Suspension
Started | 21
Completed | 19
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bimatoprost Mixed With Gonak Into a Gel Suspension
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: participants] | 46 [23 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Region of Enrollment [Number; unit: participants] — Patients were enrolled in the Bascom Palmer Eye Institute in Miami, FL.
  participants
    United States | 21
Eyelash length [Number; unit: mm] — Lash length was measured using calipers and photos during the study, and the longest measured eyelashes were plucked from the upper eyelid of 13 of the 14 total enrolled patients at the end of the six weeks for comparison. Throughout the study, we used the same measuring technique, always measuring the length of the longest lash uncurled using a surgical caliper. Visual acuity, ocular symptoms, intraocular pressure and slit lamp exam were recorded at these same intervals.
  mm
    <=18 years | 0
    Between 23 and 69 years | 21
    >69 years | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Bimatoprost in Lengthening of Eyelashes
Description: Eyelash growth after application of bimatoprost vs control (split face study).
Time Frame: 4.5 months (6 weeks of drug application and 3 months after discontinuing)
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Control Group: Each subject was given two suspensions, one of Bimatoprost mixed with Gonak into a gel suspension and one with Gonak mixed with normal saline. They were instructed to use each suspension to a pre-determined eyelash (prepared prior to study enrollment in double blind fashion and marked after randomization with right and left). The solution vials were labeled right or left eye.
Arm/Group | Bimatoprost Mixed With Gonak Into a Gel Suspension | Control Group
Number analyzed (Participants) | 19 | 19
mm | 2 (0.001) | 1.1 (0.001)

ADVERSE EVENTS:
Time Frame: 4.5 months
Description: Serious adverse events = 0 Minor adverse events (irritation) = 2 subjects, discontinued from the study. It was not documented if the adverse events were only seen in the eye with the treatment arm and thus it was documented by subjects.
Arm/Group | Bimatoprost Mixed With Gonak Into a Gel Suspension
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 2/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bimatoprost Mixed With Gonak Into a Gel Suspension (N=21)
Minor Irritation (Eye disorders) | 2 (2) — Minor irritation, conjunctival injection

LIMITATIONS AND CAVEATS:
A larger and longer term study would help assess the incidence of ocular side effects related to the Bimatoprost. This randomized controlled study evaluated patients after only 6 weeks of application of the drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes